CLINICAL TRIAL: NCT06731647
Title: Non-steroidal Anti-inflammatory Drugs in Pleurodesis Surgery for Pneumothorax
Brief Title: Non-steroidal Anti-inflammatory Drugs in Pleurodesis
Acronym: KETOTHORAX
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Collaborators: Centre Hospitalier VALENCIENNES (Other); Clinique Victor Pauchet (Other); University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PI2021_843_0175
Record Dates: First submitted 2024-12-04; First posted 2024-12-12 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2024-12

CONDITIONS: Non-steroidal Anti-inflammatory Drugs; Pleurodesis; Pneumothorax; Pain Management
Keywords: non-steroidal anti-inflammatory drugs; pleurodesis; pneumothorax; pain management
MeSH Terms: conditions — Pneumothorax; Agnosia

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Interventional group (Experimental): one intravenous dose of ketoprofen 100 mg followed by 5 doses every 12 h of ketoprofen LP 100 mg (a total regimen of 6 doses of ketoprofen every 12 h for 72h)
  Interventions: Procedure: pleurodesis procedures; Drug: KETOPROFEN(RP19583)
- Control group (Placebo Comparator): placebo of ketoprofen with the schema of administration consisting in the administration of one intravenous dose of 100 ml of NaCl 0.9% following 6 oral intakes of a placebo pill every 12h (a total regimen of 6 doses of placebo of NSAID every 12 h for 72h)
  Interventions: Procedure: pleurodesis procedures; Drug: Placebo

INTERVENTIONS:
Procedure: pleurodesis procedures — All pleurodesis procedures will be conducted with a general anesthesia. The choice of hypnotic, analgesic and neuromuscular drugs will be at the discretion of the physician. Selective orotracheal intubation will be done for all patients with a double lumen tube or a blocker according to centers habits. Regional anesthesia (serratus block, paravertebral block and erector spinae block) will be allowed and chosen at the discretion of the physician. Multimodal pain management will be allowed with the use dexamethasone, ketamine and antinociceptive drugs (nefopam, tramadol, paracetamol at the discretion of the physician. After the surgical procedure, the pleural production of liquid or air will be monitored with a chest tube connected to pleural drainage device according to centers habits. Pain will be monitored with during the hospital stay every 12 h using the pain rate scale graded from 0 to 10. Neuropathic pain will be screened at 48h, 1 months, 6 months and 1 year after the inclusion
Drug: KETOPROFEN(RP19583) — one intravenous dose of ketoprofen 100 mg followed by 5 doses every 12 h of ketoprofen LP 100 mg (a total regimen of 6 doses of ketoprofen every 12 h for 72h)
  Arms: Interventional group
Drug: Placebo — placebo of ketoprofen with the schema of administration consisting in the administration of one intravenous dose of 100 ml of NaCl 0.9% following 6 oral intakes of a placebo pill every 12h (a total regimen of 6 doses of placebo of NSAID every 12 h for 72h)
  Arms: Control group

SUMMARY:
Non-steroidal anti-inflammatory drugs (NSAIDs) are recommended in a multimodal pain management to reduce pain intensity and to spare opioid use. However, there is a controversy in its use in pleurodesis surgery as it could block the process of pleurodesis in surgical pneumothorax. In addition, NSAIDs could increase the risk of pneumothorax recurrence.

The investigators hypothesized that NSAIDs are safe during pleurodesis with a better pain management without increasing the risk of pneumothorax reccurence.

ELIGIBILITY:
Inclusion Criteria:

* Age≥18-year-old
* pneumothorax with an indication of pleurodesis
* with or without minimal lung resection
* via thoracotomy or thoracoscopy

Exclusion Criteria:

* Minor patient
* Pregnant, parturient or breast-feeding patient
* Severe polytrauma (associated with the presence of a Vittel criterion)
* Purulent pleurisy
* Hemopneumothorax
* Lactose hyper sensibility
* Contraindications to NSAID
* Contraindications to tramadol
* Contraindications to paracetamol
* Curative anticoagulation
* Patients under guardians or deprived of their liberty
* Patient refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 358 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
duration of pleural drainage | from the time of orotracheal extubation to the time of pleural tube remove
  duration of pleural drainage from the time of orotracheal extubation to the time of pleural tube remove recorded in hours.

SECONDARY OUTCOMES:
postoperative pain | at 72 hours
  postoperative pain during the first 72h after surgery assessed by the numeric rating scale (NRS) every 12 h. Pain is defined by an NRS>3 out of 10
cumulative postoperative opioid equivalent dose | at 72 hours
  cumulative postoperative opioid equivalent dose (tramadol, morphine, oxycodone) recorded in milligram and during the first 72h after surgery
Postoperative pneumonia occurence | From enrollment to the end of hospital stay, up to 6 months
  Postoperative pneumonia during hospital stay
Length of hospital stay | From enrollment to the end of hospital stay, up to 6 months
  Length of hospital stay in days
homolateral or contralateral recurrence in spontaneous pneumothorax | at 1month
  Screen in homolateral or contralateral recurrence in spontaneous pneumothorax at 1month
homolateral or contralateral recurrence in spontaneous pneumothorax | at 6 months
  Screen in homolateral or contralateral recurrence in spontaneous pneumothorax at 6 months
homolateral or contralateral recurrence in spontaneous pneumothorax | at 12 months
  Screen in homolateral or contralateral recurrence in spontaneous pneumothorax at 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Universitaire d'Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No